CLINICAL TRIAL: NCT06141226
Title: Randomized, Double-blind, Parallel Controlled, Multicenter Phase II Clinical Trial to Evaluate the Safety and Efficacy of TQB2450 Injection Combined With Arotinib Capsules and Chemotherapy in the Treatment of Advanced Non-small Cell Lung Cancer After Immune Resistance
Brief Title: Phase II Clinical Trial to Evaluate the Safety and Efficacy of TQB2450 Injection Combined With Anlotinib Capsule and Chemotherapy in the Treatment of Immunoresistant Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB2450-ALTN-II-02
Record Dates: First submitted 2023-11-14; First posted 2023-11-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 +Anlotinib+Docetaxel (Experimental): TQB2450（1200mg intravenous(iv). 3 weeks using a(q3w), day 1(d1)）+Anlotinib administered PO at day 1-14 every 3 weeks+Docetaxel（60mg/square meter intravenous(iv). 3 weeks using a(q3w), day 1(d1)）
  Interventions: Drug: TQB2450 +Anlotinib+Docetaxel
- TQB2450 +Androtinib Placebo+Docetaxel (Placebo Comparator): TQB2450 Injection（1200mg intravenous(iv). 3 weeks using a(q3w), day 1(d1)）+Anlotinib capsule placebo administered PO at day 1-14 every 3 weeks+Docetaxel Injection（60mg/square meter intravenous(iv),q3w, d1）
  Interventions: Drug: TQB2450 +Androtinib Placebo+Docetaxel

INTERVENTIONS:
Drug: TQB2450 +Anlotinib+Docetaxel — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand 1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on the surface of T cells, restoring T cell activity and enhancing immune response. It has the potential to treat various types of tumors.
  Anlotinib is a multi target receptor tyrosine kinase (RTK) inhibitor. It can inhibit VEGFR1, VEGFR2, VEGFR3, c-Kit, PDGFR β Activity.
  Docetaxel is a taxane based anti-tumor drug.
  Other Names: TQB2450/Anlotinib/Docetaxel
  Arms: TQB2450 +Anlotinib+Docetaxel
Drug: TQB2450 +Androtinib Placebo+Docetaxel — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand 1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on the surface of T cells, restoring T cell activity and enhancing immune response. It has the potential to treat various types of tumors.
  Androtinib Placebo Docetaxel is a taxane based anti-tumor drug.
  Other Names: TQB2450/Anlotinib Placebo/Docetaxel
  Arms: TQB2450 +Androtinib Placebo+Docetaxel

SUMMARY:
Objective to compare the efficacy and safety of TQB2450 injection combined with anlotinib and chemotherapy, and TQB2450 injection combined with chemotherapy in the treatment of advanced non-small cell lung cancer subjects who failed to receive first-line chemotherapy combined with immunization, and to explore and evaluate biomarkers related to efficacy, mechanism of action / resistance mechanism, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. According to the International Association for the Study of Lung Cancer and the Joint Committee on the American Classification of Cancer, 8th edition TNM staging of lung cancer, patients with locally advanced (stage IIIB/IIIC), metastatic or recurrent (stage IV) NSCLC who are histologically proven to be inoperable and unable to undergo radical synchronous radiotherapy and chemotherapy.
2. 18 years old ≤ age ≤ 75 years old; No gender limit; ECOG score 0-1 points; The expected survival period is ≥ 3 months.
3. According to RECIST 1.1 standard, there should be at least one measurable lesion.
4. Tumor resistance has progressed after receiving first-line treatment with immune checkpoint inhibitors (including PD-1 or PD-L1 monoclonal or dual antibodies) combined with platinum based drugs in the past. For neoadjuvant/adjuvant chemotherapy or radiotherapy or concurrent radiotherapy and chemotherapy, if the disease progresses during treatment or within 6 months after discontinuation of treatment, it should be considered as a first-line treatment plan.
5. It is necessary to provide tumor tissue sections that have been diagnosed with advanced or metastatic NSCLC and have not undergone radiotherapy (at least 5 samples are required for PD-L1 testing of tumor tissue, but if testing has been conducted before the first line treatment, recognized test results from each participating center can be accepted.) Tumor tissue samples must be archived samples or freshly obtained samples within the first 12 months of randomization.
6. Except for patients with squamous NSCLC, enrolled patients need to demonstrate the absence of EGFR gene sensitive mutations, ALK fusion oncogenes, or ROS1 fusion oncogenes. If it is adenosquamous cell carcinoma, stratification needs to be determined based on the dominant tissue composition.
7. Good function of main organs
8. Women of childbearing age should agree to use effective contraceptive measures during the study period and within 6 months after the end of the study. Serum pregnancy or urine pregnancy tests should be negative within 7 days before enrollment in the study; Men should agree to use effective contraceptive measures during the study period and within 6 months after the end of the study period.
9. The subjects voluntarily joined this study, signed an informed consent form, and had good compliance.

   Exclusion Criteria:
   1. Tumor diseases and medical history:

      a) If there is a central nervous system metastasis before enrollment, enrollment can be made if all the following criteria are met: i. Previously received brain metastasis treatment and met all of the following criteria:

      ① Only supratentorial and cerebellar metastases are allowed (i.e. transfer to the midbrain, pons, medulla, or spinal cord is not allowed);

      ② No imaging evidence of new or enlarged brain metastases was found;

      ③ There are no symptoms of brain metastasis, and the subject must have stopped using corticosteroids/dehydrating agents for at least 2 weeks before starting to use the investigational drug.

      Ii. Has not received brain metastasis treatment in the past and meets all of the following criteria:
      * No more than 3 metastatic lesions; ② The total length and diameter of all lesions ≤ 1.5cm;

        * There are no neurological symptoms caused by brain tissue compression;

          ④ Before starting to use the investigational drug, the subject must have stopped using corticosteroids/dehydrating agents for at least 2 weeks.

          b) There were no active malignant tumors for ≤ 2 years before randomization. c) Central type squamous cell carcinoma with a cavity (primary in the main bronchus and around the hilum of the lungs).

          d) Imaging shows that the tumor invades large blood vessels, or the boundary between the tumor and the blood vessels is unclear, or the researcher determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies.

          e) (1) Severe bone damage caused by tumor bone metastasis, including pathological fractures of load-bearing bones (such as spinal vertebrae, pelvis, femur, tibia, phalanges, calcaneus, etc.) and spinal cord compression that occur within 6 months; (2) Imaging examination suggests the presence of three or more multiple bone metastases in the load-bearing bone.

          f) Patients with serous cavity (pleural, abdominal, or pericardial) effusion that requires repeated drainage to alleviate clinical symptoms (as determined by the researcher), or those who have received serous cavity effusion drainage for treatment purposes within 2 weeks prior to treatment.
   2. Previous anti-tumor treatment:

      1. Within 2 weeks before the start of the study treatment, he received traditional Chinese patent medicines and simple preparations with anti-tumor indications specified in the NMPA approved drug instructions.
      2. I have previously used anti angiogenic drug systems such as arotinib, apatinib, lenvatinib, sorafenib, sunitinib, regofinib, and furoquitinib to treat locally advanced or metastatic NSCLC.
      3. Previously received docetaxel for systematic treatment of locally advanced or metastatic NSCLC.
      4. Unacceptable toxicity after previous anti PD - (L) 1 treatment.
      5. Patients who have received medication with immunomodulatory effects within 30 days before starting treatment.
      6. Before randomization, there are any symptoms that require systemic treatment with corticosteroids (prednisone or equivalent doses of similar drugs above 10 mg/d) or other immunosuppressive agents for ≤ 14 days.
      7. Failure to recover from toxicity and/or complications of previous intervention measures to CTCAE ≤ 1 level, except for peripheral neuropathy with hair loss and ≤ 2 level.
   3. Concomitant diseases and medical history:

      a) Decompensated cirrhosis (Child Pugh liver function rating B or C), active hepatitis, and active COVID-19 infection.

      b) Renal abnormalities: i. Renal failure requires hemodialysis or peritoneal dialysis; Ii. Previous or existing nephrotic syndrome (excluding cured), chronic nephritis.

      c) Cardiovascular and cerebrovascular abnormalities: d) Gastrointestinal abnormalities: i. Inability to take medication orally; Ii. History of malabsorption syndrome or other diseases that can interfere with gastrointestinal absorption, including a history of partial surgical removal of the stomach or intestines (excluding appendectomy); Iii. Received treatment for active gastrointestinal ulcers within the past 6 months.

      e) History of Immunodeficiency: i. Having a history of immunodeficiency, including HIV positive or suffering from other acquired or congenital immunodeficiency diseases; Ii. A history of active autoimmune diseases or autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, autoimmune hepatitis/enteritis/vasculitis/nephritis, etc; Iii. Prepare to undergo or have previously received organ transplantation; f) Bleeding risk: i. Suffering from bleeding, coagulation disorders, or using warfarin, aspirin, and other antiplatelet agglutination drugs within 28 days prior to the start of treatment (excluding preventive medication with aspirin ≤ 100 mg/d); Ii. Have a history of hemoptysis within 28 days before the start of treatment; Iii. Regardless of the severity, patients with congenital bleeding or coagulation disorders, or those who are currently using anticoagulants for treatment; Iv. Major surgical treatment or obvious traumatic injury received within 28 days prior to the start of the study treatment; v. Long term uncured wounds or fractures, excluding pathological fractures. g) Type I diabetes or II diabetes is poorly controlled. h) Having experienced severe infection of level 4 or higher within one year prior to the start of the study treatment; Subjects with 2-3 levels of active infection within 2 weeks prior to the start of study treatment; Treponema pallidum antibody (TP Ab) positive; Or those who experience unexplained fever of>38.0 ℃ during the screening period or before the first administration, or who require medical intervention.

      i) Previous or existing pneumoconiosis, interstitial pneumonia, non infectious pneumonia requiring corticosteroid treatment, currently suffering from grade 2 or other types of pneumonia, or objective evidence of severe impairment of lung function confirmed by pulmonary function examination (FEV1 or DLCO or DLCO/VA accounting for% of expected value<40%).

      j) Patients with active tuberculosis within one year prior to enrollment. k) Allergic constitution, or a history of severe allergies, or severe hypersensitivity reactions after receiving other monoclonal antibody treatments, or known allergies to the study drug excipients, or allergies to Tween 80.

      l) Previous history of severe mental disorders. m) Individuals with a history of drug abuse, alcohol or drug abuse.
   4. The end of previous clinical studies (last administration) is less than 4 weeks or the 5 half-lives of the study drug, whichever is shorter.
   5. Vaccination history within the first 28 days of randomization or vaccination during the planned study period.
   6. Pregnant or lactating female patients.
   7. According to the researcher's viewpoint, it may increase the risk associated with participating in the study, or other reasons may make it unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 48 weeks
  PFS will be defined as median number of months from the date of randomization until the first documented sign of disease progression or death due to any causes, whichever occurs first.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 48 weeks
  Objective response rate refers to the percentage of complete response (CR) or partial response (PR) subjects determined by the investigator based on Response Evaluation Criteria in Solid Tumors(RECIST) 1.1 or modified RECIST1.1 for immune based therapeutics(iRECIST) (CR and PR under iRECIST criteria can occur after imaging disease progression).
Disease control rate（DCR） | up to 48 weeks
  Disease control rate refers to the percentage of subjects with CR, PR, or stable disease (SD) of 6 weeks or more as determined by RECIST 1.1 or iRECIST (CR, PR, SD under iRECIST criteria can occur after imaging disease progression).
Overall survival (OS) | Baseline up to die
  Overall survival defined as the time from enrollment to death from any cause.
Duration of Response (DOR) | up to 48 weeks
  DOR will be defined as median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Central People's Hospital of Huizhou, Huizhou, Guangdong
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Weihai Municipal Hospital, Weihai, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality